CLINICAL TRIAL: NCT03452111
Title: Clinical Evaluation of Daily Application of Nestorone® (NES) and Testosterone (T) Combination Gel for Male Contraception
Brief Title: Study of Daily Application of Nestorone® (NES) and Testosterone (T) Combination Gel for Male Contraception
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Population Council (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kimberly Myer, Senior Program Director, NICHD, Premier Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCN017
Record Dates: First submitted 2018-02-23; First posted 2018-03-02 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Healthy; Men; Male Contraception
Keywords: Healthy Men; Couple; Gel; Male Contraception; Nestorone; Testosterone
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — ST 1435

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nestorone (NES) + testosterone (T) combined gel (Experimental): A combination Gel with Nestorone® (NES) and Testosterone (T) applied transdermally (NES/T gel). The amount of gel to be applied daily will be approximately 5 mL in volume (2.5 mL to each shoulder and upper arm per day). This daily gel volume will contain approximately 62 mg or 74 mg of T of which 6.2 mg of T with the original dose (Cohort A) and about 7.4mg of T with the second dose (Cohort B) will be absorbed per day (10% skin absorption)
  Interventions: Drug: Nestorone + Testosterone Combination Gel

INTERVENTIONS:
Drug: Nestorone + Testosterone Combination Gel — The combined gel is a transdermal treatment that will be applied daily for 52 weeks to a male subject's arms and shoulders. The formulation will be a hydro alcoholic gel. About 9 to 14% of the steroid (T or NES) in the gel applied is available to the body. The amount of gel to be applied each application will be approximately 5 mL in volume.
  Other Names: NES/T gel

SUMMARY:
The long term objective is to develop a gel to be used as a male contraceptive.

DETAILED DESCRIPTION:
This is a prospective, phase IIb, open label, single arm, multicenter study. The study protocol consists of a screening phase lasting 4 to 8 weeks, a suppression phase estimated up to 20 weeks, a 52-week maintenance/efficacy phase, and a 24-week (estimated) recovery phase.

The study will involve approximately 420 couples recruited throughout the CCTN that meet eligibility criteria. Approximately fifteen sites propose to enroll up to 420 couples (about 30 to 60 couples per site) with a goal of obtaining 200 couples completing the contraceptive efficacy phase of the study. The study has four phases (screening phase, suppression phase, efficacy phase and recovery phase) with monthly visits to provide the male participants with the NES/T gel, to encourage adherence, to monitor for possible side effects, and to quantify semen parameters. The female partner will be contacted monthly and come in for a visit every three months. Male subjects will be treated and followed as outpatients, along with their participating female partner.

ELIGIBILITY:
Inclusion Male participant - Inclusion Criteria

Men who meet all the following criteria will be eligible for enrollment in the trial:

1. Good health as confirmed by medical history, physical examination, and clinical laboratory tests of blood and urine at the time of screening;
2. 18 to 50 years of age, at the enrollment visit;
3. BMI < 33 kg/m2;
4. No history of androgen use in the six months prior to the first screening visit;
5. Agreement to use an effective method of contraception with his female partner (refer to Appendix 11 for acceptable forms of contraception) during the suppression and the first 7 days of the recovery phase and then only use the experimental method during the efficacy phase of the study;
6. In the opinion of the investigator, the male subject is willing and able to comply with the protocol, understand and sign an informed consent and HIPAA form;
7. The subject is legally competent, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions and has duly signed the informed consent form (ICF);
8. Sexually active with a female partner (as specified below) with whom he has been in a stable, mutually monogamous relationship for at least 1 year prior to screening and with whom he intends to remain in a relationship for the duration of the study;
9. No known infertility;
10. Normal reproductive state as demonstrated by:

    * Sperm concentration ≥15 million/mL in two semen samples and with no gross abnormalities of sperm motility and morphology on at least one semen sample assessment;
    * Screening Testosterone within the study site's local lab normal reference range for adult men;
11. Willingness to accept a low but unknown risk of conceiving a pregnancy for the duration of the trial.

Female participant - Inclusion Criteria

Women who meet all the following criteria will be eligible for enrollment in the trial:

1. Good general health with no chronic medical conditions that result in periodic exacerbations which require significant medical care or are known to affect fertility;
2. Aged between 18 and 34 years, inclusive, at the enrollment visit;
3. Have regular menstrual cycles of 21-35 days in duration, per patient report, when not using hormonal contraception. If hormonal contraception has been used, the following applies:

   1. If recently used intramuscular Depo-Provera must have had last injection at least 3 months prior enrollment;
   2. If using an IUD or an implant, she is planning to have this removed for purposes unrelated to enrollment in the study prior to entering the efficacy phase;
   3. Completion of her last pack of oral contraceptives or completion of effectiveness period for a monthly injection, patch or ring if any has been used prior to entering the efficacy phase;
4. Have intact uterus and at least one ovary;
5. The subject is legally competent, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions and has duly signed the informed consent form (ICF);
6. Consistent use of effective contraception during the preceding cycle prior to enrolling;
7. No known infertility;
8. Intends to remain in a monogamous relationship with male study partner (as specified above). (Note: this study will not provide her contraception for intercourse with any other male partners);
9. Be at risk for pregnancy with participating male partner (heterosexual vaginal intercourse at least once per cycle and not sterilized);
10. Have a negative pregnancy test at enrollment;
11. Willingness to accept a low but unknown risk of pregnancy and able to understand the need for follow-up in case of pregnancy;
12. No medical contraindication to pregnancy;

Exclusion Male participant - Exclusion Criteria

Men who meet any of the following criteria are not eligible for enrollment in the trial:

1. Men participating in another clinical trial involving an investigational drug within the last 30 days (or within five half-lives of the investigational drug, whichever is longer) prior to the first screening visit.
2. Men not living in the catchment's area of the study site or within a reasonable distance from the site.
3. Clinically significant abnormal findings at screening per the Investigator's medical judgment.
4. Elevated PSA levels ≥ 4 ng/mL.
5. Abnormal serum chemistry values that may indicate clinically significant liver or kidney dysfunction.
6. Use of androgens or other anabolic steroids that may suppress gonadotropins within 6 months prior to the first screening visit.
7. Diastolic blood pressure (DBP) ≥ 85 and Systolic blood pressure (SBP) ≥ 135 mm Hg; (BP will be taken three times at approximately 5 minute intervals and the mean of the 2 measurements will be used to determine eligibility).
8. History of hypertension, including hypertension controlled with treatment.
9. Known history of primary testicular disease or disorders of the hypothalamic-pituitary axis.
10. Known hypersensitivity to progestins or testosterone or any excipient of the investigational product.
11. History of prostate, testicular or breast carcinoma.
12. Significant prostatic symptoms (IPSS > 15).
13. Known history of reproductive dysfunction including vasectomy or infertility.
14. Known history of significant cardiac, renal, hepatic or prostatic disease.
15. History of thromboembolic disease.
16. A serious systemic disease such as diabetes mellitus (including diabetes controlled with treatment), HIV/AIDS;
17. Current active or ongoing Hepatitis infection.
18. History of untreated sleep apnea.
19. Known or suspected current alcohol dependence syndrome, chronic marijuana use, or any illicit drug use that may affect metabolism/transformation of steroid hormones and study treatment compliance.
20. Any skin condition that might interfere with absorption of gel.
21. Couples desiring fertility within the study participation period (approximately 104 weeks from screening to end of recovery).
22. PHQ9 score ≥10, a score ≥1 on Question #9 on the PHQ9, or history of severe depression or other serious mental health disorder, including ongoing use of an anti-depressant.
23. Men participating in competitive sports where drug screening for prohibited substances (including anabolic steroids) is routine. Exclusion is due to the potential of testing positive for androgens that may occur from their study participation coupled with the unknown efficacy (i.e. duration of positive testing) of a single application.
24. Use of sex steroids or medications which might interfere with steroid metabolism (i.e., ketoconazole, finasteride, oral corticosteroids, dutasteride, and statins).
25. Use of anticoagulants.
26. Use of medications that will interfere or interact with Nestorone or Testosterone.
27. Use of oily cosmetic skin gels/products that would prevent absorption of steroids.
28. Previous participation in this clinical trial.
29. Any site staff member with delegated study responsibilities or a family member of a site staff member with delegated study responsibilities.
30. Have issues or concerns (in the judgment of the investigator) that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study.

Female participant - Exclusion Criteria

1. Desire to become pregnant during the study.
2. Breastfeeding.
3. Known or suspected current alcoholism or drug abuse.
4. Participation in another clinical trial involving an investigational drug within the last 30 days prior to the first screening visit.
5. Currently pregnant.
6. Known hypersensitivity to progestins or testosterone.
7. Previous participation in this clinical trial.
8. Any site staff member with delegated study responsibilities or a family member of a site staff member with delegated study responsibilities.
9. Have issues or concerns (in the judgment of the investigator) that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 420 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Contraceptive efficacy provided by daily application of NES/T gel for 52 wks during the efficacy phase of the study determined using Kaplan-Meier methods to estimate the 12-mth cumulative pregnancy probability in the efficacy(evaluable cycles)population. | 12 months

SECONDARY OUTCOMES:
Suppression of spermatogenesis induced by daily use of the NES/T gel as assessed by semen analyses using number of subjects with sperm concentration <1 million (M)/mL during the suppression phase of the study. | 20 weeks
Maintenance of suppression of spermatogensis induced by daily use of the NES/T gel as assessed by semen analyses using number of subjects with sperm concentration <1 million (M)/mL during the 52 week efficacy phase of the study. | 52 weeks
Changes from baseline in Follicle Stimulating Hormone (FSH) with daily use of the NES/T gel. | 24 months
Changes from baseline in Luteinizing Hormone (LH) with daily use of the NES/T gel. | 24 months
Changes from baseline in Sex Hormone Binding Globulin (SHBG) with daily use of the NES/T gel. | 24 months
Changes from baseline in Testosterone with daily use of the NES/T gel. | 24 months
Changes from baseline in Nestorone with daily use of the NES/T gel. | 24 months
Incidence of treatment emergent adverse events with daily use of the NES/T gel. | 24 months
Changes from baseline in sodium with daily use of the NES/T gel. | 24 months
Changes from baseline in potassium with daily use of the NES/T gel. | 24 months
Changes from baseline in chloride with daily use of the NES/T gel. | 24 months
Changes from baseline in bicarbonate with daily use of the NES/T gel. | 24 months
Changes from baseline in fasting glucose with daily use of the NES/T gel. | 24 months
Changes from baseline in blood urea nitrogen with daily use of the NES/T gel. | 24 months
Changes from baseline in creatinine with daily use of the NES/T gel. | 24 months
Changes from baseline in calcium with daily use of the NES/T gel. | 24 months
Changes from baseline in total bilirubin with daily use of the NES/T gel. | 24 months
Changes from baseline in alkaline phosphatase with daily use of the NES/T gel. | 24 months
Changes from baseline in alanine aminotransferase with daily use of the NES/T gel. | 24 months
Changes from baseline in aspartate transaminase with daily use of the NES/T gel. | 24 months
Changes from baseline in albumin with daily use of the NES/T gel. | 24 months
Changes from baseline in mood with daily use of the NES/T gel using the Patient Health Questionnaire-9. | 24 months
Changes from baseline in sexual function with daily use of the NES/T gel using the psychosexual daily questionnaire. | 24 months
Changes from baseline in prostate function with daily use of NES/T gel using the International Prostate Symptom Score. | 24 months
Acceptability of NES/T gel as a contraceptive among male and female participants using the acceptability questionnaires. | 24 months
Length of time to recovery of spermatogenesis after daily use of NES/T gel as assessed by sperm concentration > 15 million (M)/mL during the recovery phase. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diana Blithe, PhD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (17):
- United States (9):
  - UC Davis Health, Sacramento, California
  - The Lunquist Institute at Harbor-UCLA Medical Center, Torrance, California
  - Comprehensive Women's Health Center, Denver, Colorado
  - University of Kansas, Kansas City, Kansas
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Eastern Virginia Medical School-EVMS Obstetrics & Gynecology, Norfolk, Virginia
  - University of Washington Medical Center & Health Sciences, Seattle, Washington
- Chile (2):
  - Centro de Medicina Reproductiva Shady Grove Chile, Santiago, Vitacura
  - Chilean Institute of Reproductive Medicine, Santiago
- University of Bologna, Italy, Bologna, Italy
- Kenyatta National Hospital, Nairobi, Kenya
- Karolinska Institutet, Stockholm, Sweden
- United Kingdom (2):
  - University of Edinburgh, Edinburgh
  - University of Manchester, UK, Manchester
- Spilhaus Clinical Research Site, Harare, Zimbabwe

REFERENCES:
- [Derived] Lue Y, Swerdloff R, Pak Y, Nguyen BT, Yuen F, Liu PY, Blithe DL, Wang C. Male contraception development: monitoring effective spermatogenesis suppression utilizing a user-controlled sperm concentration test compared with standard semen analysis. Fertil Steril. 2023 Feb;119(2):208-217. doi: 10.1016/j.fertnstert.2022.11.002. Epub 2022 Nov 5. PMID 36347310